CLINICAL TRIAL: NCT02375230
Title: MRSOPA-Drills to Improve Mask Ventilation in the Delivery Room
Acronym: MRSOPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00054147
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Apnea; Bradycardia
Keywords: Neonatal Resuscitation; Respiratory Function Tests; Neonatal Simulation; Resuscitation Teaching
MeSH Terms: conditions — Apnea; Bradycardia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): "Control group"
  Health care provider randomized to the control group will receive a copy of the NRP text pages discussing MR SOPA at every shift for self-study. They will be encouraged by the educator to study these pages for five minutes at every shift. The educator will be there to answer questions if they arise.
  Interventions: Procedure: Control group
- MR SOPA (Active Comparator): Health care provider randomized to the "MR SOPA" group will receive MR SOPA training provided by a qualified educator on every shift. This training will be five minutes long and will consist of each MR SOPA step. These corrective steps will be demonstrated and practiced on a low-fidelity neonatal mannequin. Each participant will receive five minutes of training at the start of each shift.
  The educator will teach mask adjustment, and airway reposition. If either of these first steps is unsuccessful the participant will learn about mouth and nose suction, open mouth and increase of airway pressure. All participants will also learn and practice alternative airways placement including intubation and laryngeal mask airway placement.
  Interventions: Procedure: MR SOPA

INTERVENTIONS:
Procedure: Control group — Health care provider randomized to the control group will receive a copy of the NRP text pages discussing MR SOPA at every shift for self-study. They will be encouraged by the educator to study these pages for five minutes at every shift. The educator will be there to answer questions if they arise.
  Arms: Control
Procedure: MR SOPA — Health care provider randomized to the "MR SOPA" group will receive MR SOPA training provided by a qualified educator on every shift. This training will be five minutes long and will consist of each MR SOPA step. These corrective steps will be demonstrated and practiced on a low-fidelity neonatal mannequin. The alternative airway practice will be performed on an intubation mannequin in the DR also placed on the DR resuscitation unit. Each participant will receive five minutes of training at the start of each shift.
  Arms: MR SOPA

SUMMARY:
Establishing breathing after birth is vital for survival and long-term health of premature babies. 10% of all preterm babies fail to breathe after birth and require help with breathing. When infants need help with breathing the clinical team will place a small mask on the babies face to give some breaths to help the baby breath (what the investigators call mask ventilation).

This procedure is done million times a day around the world and several times a day here at the Royal Alexandra Hospital. Providing these breaths via mask ventilation is the most difficult step in helping a baby breath at birth. If this is provided wrongly then baby does not receive enough oxygen, which could damage the brain and even cause death.

To keep the skill level of every staff member up-to-date every staff member is required to re-train this rescue breaths via mask ventilation once every two years.

The investigators believe this is not enough and that daily trainings are necessary to keep your skills up-to-date.

The investigators aim to compare to different teaching techniques using daily trainings to see if either improves the skills of the resuscitator providing mask ventilation

The study will last 7 month (baseline observations (2 months), intervention period (3 months), After trial period (2 months)

The investigators will use our routinely used equipment to record neonatal resuscitation and the investigators also routinely make video recordings to evaluate performance during resuscitation.

DETAILED DESCRIPTION:
Background

Establishing breathing and oxygenation after birth is vital for survival and long-term health of premature infants. 10% of all preterm infants fail to breathe after birth and require respiratory support. An international consensus statement recommends that infants with inadequate breathing or bradycardia after birth be given positive pressure ventilation (PPV) via a facemask with a T-piece device. Mannequin and DR studies have shown that PPV is difficult and mask leak and airway obstruction are common problems during PPV. Several factors such as poor facemask application resulting in leak or airway obstruction, spontaneous movements of the baby, movements by or distraction of the resuscitator, changing the wet towels or putting a hat can reduce the effectiveness of PPV. We recently reported both that significant airway obstruction and mask leaks occur in about half of the very preterm infants who received PPV in the DR. In particular, large mask leak was observed in twice as many recordings as airway obstruction and only in about a third of recordings neither obstruction nor facemask leak occurred. In addition, mask leak was more likely to occur at the start of PPV, while airway obstruction more often occurred later on. Assessment of the infant may distract the resuscitators focus from mask position and mask holding techniques during the initial phase of PPV.

MR SOPA

Neonatal Resuscitation Program (NRP) emphasizes on the ventilation corrective steps to ensure effective mask ventilation before moving to the next steps of resuscitation. Technique for improving PPV by mask is performed by a series of corrective steps, identified by the acronym "MR SOPA", to recall ventilation corrective steps. The steps should be followed with this order: "M Mask adjustment, R Reposition airway, S Suction mouth and nose, O Open mouth, P Pressure increase, A Airway alternative".

Hypotheses to be tested

We hypothesize that improved mask ventilation techniques using daily MRSOPA-Drills (MR SOPA group) compared to standard NRP teaching (control group) will reduce mask leak in preterm infants <33 weeks gestation who requiring breathing support at birth. We aim to determine if daily MR SOPA Drills compared to standard NRP teaching improves mask ventilation.

Experimental design and methods

Study population: Infants <33 weeks gestation requiring respiratory support at birth will be included if member of the Resuscitation-Stabilization-Triage team (RST-team) enrolled in study attend deliveries.

Study design: Randomized controlled trial.

Participants: Members of the RST-team, which usually consists of a neonatal nurse (n=50), neonatal respiratory therapist (n=30), neonatal nurse practitioner (n=16) or neonatal fellow (n=6), and a neonatal consultant (n=15). Deliveries are usually attended by a minimum of three RST-Team members: a neonatal nurse, neonatal respiratory therapist and neonatal nurse practitioner or neonatal fellow. Participants of each professional group will be randomized after informed consent and members of each professional group will be stratified to both groups.

In addition, should state that babies health information will be collected

Description of interventions and timeline

Interventions for both groups ("MR SOPA group" and "control group")

Baseline (2 months)

Over a period of two months all participants will be recorded during several real-life resuscitations using our unique recording system (including respiratory function monitoring and video recordings) to establish a baseline of mask PPV performance.

Intervention period

"MR SOPA group"

Health care provider randomized to the "MR SOPA" group will receive MR SOPA training provided by a qualified educator on every shift. This training will be five minutes long and will consist of each MR SOPA step. These corrective steps will be demonstrated and practiced on a low-fidelity neonatal mannequin in the DR of the Royal Alexandra Hospital. The mannequin will be placed on our DR resuscitation unit to simulate real-life scenarios. The alternative airway practice will be performed on an intubation mannequin in the DR also placed on the DR resuscitation unit. Each participant will receive five minutes of training at the start of each shift.

The educator will teach mask adjustment, and airway reposition. If either of these first steps is unsuccessful the participant will learn about mouth and nose suction, open mouth and increase of airway pressure. All participants will also learn and practice alternative airways placement including intubation and laryngeal mask airway placement.

"Control group"

Health care provider randomized to the control group will receive a copy of the NRP text pages discussing MR SOPA at every shift for self-study. They will be encouraged by the educator to study these pages for five minutes at every shift. The educator will be there to answer questions if they arise.

After trial period (2 months)

After recruiting and training the study participants in the intervention period the real life resuscitations will be recorded similarly as in the pre-trial period over the next two months, using our unique recording system. This period will be compared to the baselines measures in the pre-trial period.

Resuscitation

All resuscitative measures will be decided by the RST-team, in accordance with the 2010 guidelines for neonatal resuscitation.

Equipment for recording resuscitations

We will use our routinely used equipment to record neonatal resuscitation including a user-friendly respiratory function monitor will measure respiratory parameters including tidal volume, airway pressures, gas flow, minute ventilation, and exhaled CO2. Percutaneous oxygen saturation will be assessed using pulse oximetery and systemic and regional hemodynamic function will be assessed using heart rate, and blood pressure. A high-definition digital video of these resuscitations will be made using a webcam.

ELIGIBILITY:
Inclusion Criteria:

* Infants <33 weeks gestation requiring respiratory support at birth will be included if member of the Resuscitation-Stabilization-Triage team (RST-team) enrolled in study attend deliveries.

Exclusion Criteria:

* Infants of parents who decline consent

Max Age: 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mask leak | within 10min after birth

SECONDARY OUTCOMES:
Rate of Intubation | within 60min after birth
Apgar score at 1min | 1min after birth
Apgar score at 5min | 5min after birth
Rate of Chest compression | within 10min after birth

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, MD,PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
data will be shared after request from researchers